CLINICAL TRIAL: NCT02319343
Title: Effect of Preoperative Intravenous High Dose Methylprednisolone on Quadriceps Muscle Function in Patients Scheduled for Total Knee-arthroplasty
Brief Title: Effect of Methylprednisolone on Quadriceps Muscle Function in Patients Undergoing Total Knee-arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Viktoria Oline Lindberg-Larsen, MD, research assistant, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: HK_VL_08_2014
Record Dates: First submitted 2014-12-08; First posted 2014-12-18 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Osteoarthrosis
Keywords: Glucocorticoid; Quadriceps muscle function; Knee arthroplasty, total
MeSH Terms: conditions — Osteoarthritis | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylprednisolone (Active Comparator): Preoperative single high dose of Solu-Medrol 125 mg iv.
  Interventions: Drug: Methylprednisolone
- Isotonic Sodium Chloride (Placebo Comparator): Preoperative single dose of isotonic Sodium Chloride.
  Interventions: Drug: Isotonic Sodium Chloride

INTERVENTIONS:
Drug: Methylprednisolone — Comparison of preoperative single high dose of Methylprednisolone 125 mg iv. and isotonic Sodium Chloride (placebo)
  Other Names: Solu-Medrol
  Arms: Methylprednisolone
Drug: Isotonic Sodium Chloride — Placebo
  Arms: Isotonic Sodium Chloride

SUMMARY:
This study evaluates the pathophysiological effects of a single dose Methylprednisolone administered prior to total knee-arthroplasty (TKA). The investigators examine the effect on thigh muscle function to evaluate the efficacy of Methylprednisolone on knee-extension strength at discharge after TKA.

Half of participants will receive intravenous Solu-Medrol 125 mg, while the other half will receive placebo.

The investigators hypothesize that the group receiving Methylprednisolone will experience smaller loss of knee-extension strength compared to the placebo-group, early after TKA.

DETAILED DESCRIPTION:
The anti-inflammatory effects of glucocorticoids are well known. The beneficial effects in postoperative pain, postoperative nausea and vomiting are well-documented.

Knee-arthroplasty surgery and the inflammatory stress response in general affect the potential of recovery. The quadriceps muscle strength is shown to be reduced significantly (80%) early after surgery. The mechanism is thought related to inhibitory reflexes and pain caused by surgical induced inflammation around the knee joint. The effect of glucocorticoids on the quadriceps muscle function after knee-arthroplasty surgery is unknown and calls for further investigation.

The study is to be considered as explorative.

The primary analysis of the primary outcome measure is a comparison of the changes in knee extension strength from baseline to 48 hours postoperatively between the two groups.

For calculation of sample size the average loss of strength from baseline (before surgery) to 48 hours after TKA-surgery being 0.8 Nm/kg body weight (SD=0.39, Holm et al. 2010), a risk of type I errors 5% and a risk of type II errors 20% (80% power) were used. The sample size is estimated to reveal a group difference in knee extension strength of minimum 40%.

The primary analysis is carried out on all included patients (intention-to-treat) with baseline values as covariate. Secondary exploratory per-protocol analysis might be performed. Missing outcomes will be analysed using multiple imputation due to expected strong time trends.

The secondary outcome measures; a group difference of 6 sec. (Timed Up & Go) and 2 cm (knee circumference) are considered clinically relevant. The statistical power is based on the calculation outlined above using the same test prerequisites.

For further details please also view the European Clinical Trials Database (EudraCT) registration:

EudraCT nr.: 2014-003395-23

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthrosis
* Undergoing total unilateral knee-arthroplasty surgery
* Speak and understand Danish
* Have given informed consent

Exclusion Criteria:

* Revision, bilateral or uni chamber knee-arthroplasty surgery
* General anaesthesia
* Allergy or intolerance towards Methylprednisolone
* Local or systemic infection
* Permanent systemic treatment with steroids within 30 days preoperatively
* Insulin-dependent diabetes
* Active treatment of ulcer within 3 months preoperatively
* Cancer disease
* Autoimmune disease incl. rheumatoid arthritis
* Pregnant or breast feeding women
* Menopause <1 year

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in isometric knee extension strength measured as Nm/kg from baseline to 48 hours after surgery | two days after surgery

SECONDARY OUTCOMES:
Change in Timed Up & Go (sec.) from baseline (before surgery) to 48 hours after surgery | two days after surgery
Change in knee circumference (cm) from baseline (before surgery) to 48 hours after surgery | two days after surgery
Change in pain intensity from baseline (before surgery) to 48 hours after surgery | two days after surgery
Change in concentration of C-reactive Protein from baseline (before surgery) to 48 hours after surgery | two days after suregry

CONTACTS AND LOCATIONS:
Overall Officials: Viktoria Lindberg-Larsen, MD, Principal Investigator — Section for Surgical Pathophysiology, Rigshospitalet
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Husted H. Fast-track hip and knee arthroplasty: clinical and organizational aspects. Acta Orthop Suppl. 2012 Oct;83(346):1-39. doi: 10.3109/17453674.2012.700593. PMID 23205862
- [Background] Kehlet H. Fast-track hip and knee arthroplasty. Lancet. 2013 May 11;381(9878):1600-2. doi: 10.1016/S0140-6736(13)61003-X. No abstract available. PMID 23663938
- [Background] Khan SK, Malviya A, Muller SD, Carluke I, Partington PF, Emmerson KP, Reed MR. Reduced short-term complications and mortality following Enhanced Recovery primary hip and knee arthroplasty: results from 6,000 consecutive procedures. Acta Orthop. 2014 Feb;85(1):26-31. doi: 10.3109/17453674.2013.874925. Epub 2013 Dec 20. PMID 24359028
- [Background] Malviya A, Martin K, Harper I, Muller SD, Emmerson KP, Partington PF, Reed MR. Enhanced recovery program for hip and knee replacement reduces death rate. Acta Orthop. 2011 Oct;82(5):577-81. doi: 10.3109/17453674.2011.618911. Epub 2011 Sep 6. PMID 21895500
- [Background] Lunn TH, Kristensen BB, Andersen LO, Husted H, Otte KS, Gaarn-Larsen L, Kehlet H. Effect of high-dose preoperative methylprednisolone on pain and recovery after total knee arthroplasty: a randomized, placebo-controlled trial. Br J Anaesth. 2011 Feb;106(2):230-8. doi: 10.1093/bja/aeq333. Epub 2010 Dec 3. PMID 21131371
- [Background] Bandholm T, Kehlet H. Physiotherapy exercise after fast-track total hip and knee arthroplasty: time for reconsideration? Arch Phys Med Rehabil. 2012 Jul;93(7):1292-4. doi: 10.1016/j.apmr.2012.02.014. Epub 2012 Feb 27. PMID 22494947
- [Background] Geborek P, Mansson B, Wollheim FA, Moritz U. Intraarticular corticosteroid injection into rheumatoid arthritis knees improves extensor muscles strength. Rheumatol Int. 1990;9(6):265-70. doi: 10.1007/BF00541322. PMID 2315606
- [Background] Rice DA, McNair PJ. Quadriceps arthrogenic muscle inhibition: neural mechanisms and treatment perspectives. Semin Arthritis Rheum. 2010 Dec;40(3):250-66. doi: 10.1016/j.semarthrit.2009.10.001. Epub 2009 Dec 2. PMID 19954822
- [Background] Holte K, Kehlet H. Perioperative single-dose glucocorticoid administration: pathophysiologic effects and clinical implications. J Am Coll Surg. 2002 Nov;195(5):694-712. doi: 10.1016/s1072-7515(02)01491-6. No abstract available. PMID 12437261
- [Result] Holm B, Kristensen MT, Bencke J, Husted H, Kehlet H, Bandholm T. Loss of knee-extension strength is related to knee swelling after total knee arthroplasty. Arch Phys Med Rehabil. 2010 Nov;91(11):1770-6. doi: 10.1016/j.apmr.2010.07.229. PMID 21044725